CLINICAL TRIAL: NCT01851525
Title: Therapeutic Outcomes Using Contact Force Handling During Atrial Fibrillation Ablation
Acronym: TOUCH AF
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Southlake Regional Health Centre (Other)
Collaborators: Applied Health Research Centre (Other)
Responsible Party: Principal Investigator, Atul Verma, Principal Investigator, Southlake Regional Health Centre
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: 01
Record Dates: First submitted 2013-05-05; First posted 2013-05-10 (Estimated); Last update posted 2017-04-25 (Actual); Status verified 2017-04

CONDITIONS: Persistent Atrial Fibrillation
Keywords: Atrial fibrillation; Ablation
MeSH Terms: conditions — Atrial Fibrillation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Contact Force Sensing (CFS) Blinded (Active Comparator): Contact Force Sensing (CFS) Blinded: Operator will be blinded to data provided by the integrated force sensor in the ablation catheter (ThermoCoolSmartTouch ablation catheter)
  Interventions: Device: ThermoCoolSmartTouch ablation catheter, Biosense Webster
- Contact Force Sensing (CFS) Guided (Active Comparator): Contact Force Sensing (CFS) Guided: Operator will be guided by integrated force sensor in the ablation catheter (ThermoCoolSmartTouch ablation catheter)
  Interventions: Device: ThermoCoolSmartTouch ablation catheter, Biosense Webster

INTERVENTIONS:
Device: ThermoCoolSmartTouch ablation catheter, Biosense Webster

SUMMARY:
Catheter ablation has emerged as an effective therapy for atrial fibrillation (AF). However, achievement of complete& durable isolation of the pulmonary veins (PVs) is challenging, primary limited both by operator experience and also the limits of currently available ablation technology. Direct contact force sensing (CFS) is a novel technology that may help to ensure adequate lesion delivery. CFS may also help to improve the safety profile of catheter ablation. The purpose of this study is to compare two strategies of wide antral PV isolation plus linear ablation for persistent AF:

1. guided by contact force sensing (CFS) OR
2. blinded to contact force sensing (CFS) - i.e. standard approach

ELIGIBILITY:
Inclusion Criteria

* Age > 18 years.
* Patients undergoing first-time catheter ablation for AF.
* Persistent AF defined as episodes greater than 7 days duration.
* Symptomatic AF defined as patients who have been aware of their AF anytime within the last 5 years prior to enrolment. Symptoms may include, but are not restricted to, palpitations, shortness of breath, chest pain, fatigue, left ventricular dysfunction, or other symptoms, or any combination of the above.
* At least one episode of AF must have been documented by ECG, Holter, loop recorder, telemetry, implanted device, or transtelephonic monitoring within 24 months of enrolment.
* Willing and able to provide informed consent.

Exclusion Criteria

* Paroxysmal AF.
* AF secondary to a reversible cause.
* Patients with contraindications to systemic anticoagulation with heparin, coumadin, or a direct thrombin inhibitor.
* Patients who have previously undergone AF ablation.
* Patients with left atrial size >55 mm (echocardiography, parasternal long axis view).
* Patients who are or may potentially be pregnant.

Min Age: 19 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 120 (Estimated)
Dates: Start 2013-06; Primary Completion 2017-02-15 (Actual); Study Completion 2017-02-15 (Actual)

PRIMARY OUTCOMES:
Total cumulative radio frequency (RF) delivery time | 12 months
  Total cumulative RF delivery time for all ablation procedures performed during the study period (12 mo)

SECONDARY OUTCOMES:
Freedom from AF or atrial arrhythmia >30 sec | 12 months
  Freedom from AF or atrial arrhythmia >30 sec at 12 months post-initial ablation
Ability to achieve PV isolation with a single ring of lesions around each PV | 6 hours
  Ability to achieve PV isolation with a single ring of lesions around each PV
Ability to achieve linear ablation with complete conduction block on the first attempt | 6 hours
  Ability to achieve linear ablation with complete conduction block on the first attempt
Number & location of conduction gaps after initial circumferential ablation lines | 6 hours
  Number & location of conduction gaps after initial circumferential ablation lines during first ablation procedure
Number & location of conduction gaps after initial linear ablation | 6 hours
  Number & location of conduction gaps after initial linear ablation during first ablation procedure
Time required for successful PV isolation | 12 months
  Time required for successful PV isolation taking into consideration all ablation procedures
Time required for successful linear ablation | 12 months
  Time required for successful linear ablation taking into consideration all ablation procedures
Total fast anatomical mapping (FAM) time | 12 months
  Total FAM time taking into consideration all ablation procedures
FAM volume | 12 months
  FAM volume of CFS vs non-CFS guided maps
Freedom from ablation-related major adverse events at 90 days post-ablation - specifically perforation, stroke/thromboembolism, esophageal injury, and symptomatic PV stenosis | 90 days
  Freedom from ablation-related major adverse events at 90 days post-ablation - specifically perforation, stroke/thromboembolism, esophageal injury, and symptomatic PV stenosis
Incidence of repeat ablation procedures | 12 months
Incidence of conduction gaps around pulmonary veins | 12 months
  Incidence of conduction gaps around pulmonary veins and correlation to force measures in those gaps
Freedom from atrial arrhythmia > 30 sec | 12 months
  Freedom from atrial arrhythmia > 30 sec at 12 months after one procedure
Freedom from atrial arrhythmia > 30 sec after one or two procedures | 12 months
  Freedom from atrial arrhythmia > 30 sec at 12 months after one or two procedures
Reduction in atrial arrhythmia burden by >90% | 12 months

CONTACTS AND LOCATIONS:
Overall Officials: Atul Verma, MD, Principal Investigator — Southlake Regional Health Centre
Locations (4):
- Canada (4):
  - Vancouver Island Cardiac Arrhythmia Clinic, Victoria, British Columbia
  - Southlake Regional Health Centre, Newmarket, Ontario
  - Montreal Heart Institute, Montreal, Quebec
  - Laval University Cardiac and Pulmonary Institute, Québec, Quebec